CLINICAL TRIAL: NCT04398238
Title: "Change in Transfusion Rates of Patients Undergoing Elective Total Hip Replacement Before/After the Implementation of a Peri-operative Patient Blood Management Program: a Retrospective Observational Study.
Brief Title: Transfusion Rates in Total Hip Replacement Before/After the Implementation of a Patient Blood Management Program.
Acronym: pbm-hip
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 346/2020/Oss/IOR
Record Dates: First submitted 2020-05-12; First posted 2020-05-21 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Anemia (Diagnosis); Iron-deficiency; Transfusion; Arthroplasty
Keywords: patient blood management; anemia; Arthroplasty
MeSH Terms: conditions — Anemia; Disease; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-PBM: patients screened for surgery before the implementation of PBM program: pre-operative evaluation and treatment according to usual care
- post-PBM: patients screened for surgery after the implementation of PBM program (3 months allowed for training/optimization): all patients with pre-operative hemoglobin < 13g/dl undergo screening for causes and treatment as needed.
  Interventions: Combination Product: evaluation by transfusion medicine specialist

INTERVENTIONS:
Combination Product: evaluation by transfusion medicine specialist — screening for anemia causes and treatment: iron/folate/vitamin B12 supplementation, Erythropoietin administration if indicated
  Groups: post-PBM

SUMMARY:
Retrospective observational study: impact of a peri-operative patient blood management program (PBM) on transfusion rates of patients undergoing elective hip replacement.

DETAILED DESCRIPTION:
A Patient Blood Management (PBM) program was implemented in year 2019 in our institution: patient scheduled for elective total hip replacement underwent pre-operative screening about one month before surgery, and those with pre-operative hemoglobin < 13 g/dl were screened for possible causes and treatment of anemia.

Data from two different time frames, before and after the implementation of the program, were collected to study the change in clinical outcomes such as transfusion rates, length of stay, etc.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective hip replacement in the selected time-frame
* American Society of Anesthesiology (ASA) status 1-2-3
* age >18

Exclusion Criteria:

* patients not undergoing screening as outpatients at pre-operative clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of age > 18 who undergo screening and surgery for hip athroplasty in the selected time-frame
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
transfusion rates | from day of surgery till day of discharge, up to 60 days
  percentage of patients undergoing hip replacement who receive at least one unit of concentrated red cells during or after surgery

SECONDARY OUTCOMES:
minimum hemoglobin | from day of surgery till day of discharge, up to 60 days
  minimum hemoglobin reached after surgery
hemoglobin at discharge | from day of surgery till day of discharge, up to 60 days
  last measured hemoglobin before discharge from hospital
length of stay | from day of surgery till day of discharge, up to 60 days
  total days of hospital stay from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bonarelli, MD, Principal Investigator — Istituto Ortopedico Rizzoli; Sandra Giannone, MD, Study Chair — Istituto Ortopedico Rizzoli
Locations (1):
- Sandra Giannone, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ellermann I, Bueckmann A, Eveslage M, Buddendick H, Latal T, Niehoff D, Geissler RG, Hempel G, Kerkhoff A, Berdel WE, Roeder N, Van Aken HK, Zarbock A, Steinbicker AU. Treating Anemia in the Preanesthesia Assessment Clinic: Results of a Retrospective Evaluation. Anesth Analg. 2018 Nov;127(5):1202-1210. doi: 10.1213/ANE.0000000000003583. PMID 29944518
- [Background] Munoz M, Acheson AG, Auerbach M, Besser M, Habler O, Kehlet H, Liumbruno GM, Lasocki S, Meybohm P, Rao Baikady R, Richards T, Shander A, So-Osman C, Spahn DR, Klein AA. International consensus statement on the peri-operative management of anaemia and iron deficiency. Anaesthesia. 2017 Feb;72(2):233-247. doi: 10.1111/anae.13773. Epub 2016 Dec 20. PMID 27996086
- [Background] Rineau E, Chaudet A, Chassier C, Bizot P, Lasocki S. Implementing a blood management protocol during the entire perioperative period allows a reduction in transfusion rate in major orthopedic surgery: a before-after study. Transfusion. 2016 Mar;56(3):673-81. doi: 10.1111/trf.13468. Epub 2016 Jan 8. PMID 26748489